CLINICAL TRIAL: NCT01571271
Title: Electrohydraulic Versus Laser Lithotripsy for Treatment of Difficult to Remove Biliary Stones
Acronym: EHLvlaser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mansour Parsi, MD, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-168; NCT01039246 (obsolete NCT alias)
Record Dates: First submitted 2009-12-23; First posted 2012-04-05 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Gall Stones
Keywords: biliary; lithotripsy; gall stones; bile duct; Biliary stones
MeSH Terms: conditions — Gallstones; Cholecystolithiasis | interventions — Lithotripsy, Laser; Lithotripsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrohydraulic lithotripsy (Experimental): Electrohydraulic lithotripsy: Lithotripsy will be performed using electrohydraulic method
  Interventions: Procedure: Electrohydraulic Lithotripsy
- Laser Lithotripsy (Experimental): Laser Lithotripsy: Lithotripsy will be performed using laser method
  Interventions: Procedure: Laser Lithotripsy

INTERVENTIONS:
Procedure: Laser Lithotripsy — Laser Lithotripsy
  Other Names: Lithotripsy
  Arms: Laser Lithotripsy
Procedure: Electrohydraulic Lithotripsy — Electrohydraulic Lithotripsy
  Arms: Electrohydraulic lithotripsy

SUMMARY:
Bile duct stones that can't be removed by conventional means can often be removed after fragmentation by shock waves (lithotripsy). The shock waves that are used for fragmentation of these stones are generated by electric sparks (electrohydraulic lithotripsy) or laser (laser lithotripsy). Although both techniques have been used for many years, there are no studies comparing the efficacy of the two. The purpose of this study is to find out which technique is more effective.

DETAILED DESCRIPTION:
Procedures will be considered standard of care; patients or insurance companies will be billed as it is standard of care.

ELIGIBILITY:
Inclusion Criteria:

* 1 or more gall stones in bile duct which cannot be removed using conventional methods (must be fragmented)
* Adults able to provide informed consent

Exclusion Criteria:

* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time | Procudre duration
  Identify which technique takes less time to completion.

SECONDARY OUTCOMES:
Number of shocks | Procedure duration
  Comparsion between procudures of the number of shocks to fragment stones

CONTACTS AND LOCATIONS:
Overall Officials: Mansour A. Parsi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No